CLINICAL TRIAL: NCT01553370
Title: Randomized Controlled Trial of Milk Products and Physical Activity on Body Composition and Health in Overweight Young Males
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, Brian Roy, Associate Professor, Brock University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BUCT-11-221
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alternate Intake-time (Active Comparator)
  Interventions: Other: Increased Dairy Intake; Other: Supplemental carbohydrate
- Immediately post-exercise (Experimental)
  Interventions: Other: Increased Dairy Intake; Other: Supplemental carbohydrate

INTERVENTIONS:
Other: Increased Dairy Intake — 3 additional servings of low fat dairy will be consumed
Other: Supplemental carbohydrate — Maltodextrin will be provided in an amount equal to the the energy content in the 3 supplemental servings of low-fat dairy.

SUMMARY:
Maintaining a healthy body weight is a major challenge for the majority of Canadians. A lifestyle strategy that promotes maintenance of a healthy body weight and, perhaps most importantly, can be incorporated into daily life with relative ease is essential. This study will determine if an effective strategy includes increased physical activity in conjunction with higher intakes of dairy products immediately following exercise. Fifty-six overweight adult males who do not regularly exercise will be assigned to one of four groups for 12 weeks. All groups will preform 12 weeks of exercise training (1 hour of cycling per day, 5 times per week). Two groups will consume supplemental low fat milk (3 servings per day) with one these groups consuming it immediately after exercise while the other will consume it either well before or long after the exercise session. The other two groups will consume a carbohydrate drink that has the same amount of energy as the low fat milk, with one of these groups consuming the drink right after exercise and the other another group will consume it either well before or long after the exercise session. Markers of health status including body weight, muscle mass, and bone mass will be measured at the start and after the 12- week intervention. The investigators anticipate that providing the low fat milk immediately after exercise will result in the most favorable changes in health outcomes, and provide a realistic lifestyle intervention for overweight individuals to attain a healthy body weight, and by doing so, optimize their ability to prevent chronic disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater or equal to 25
* healthy

Exclusion Criteria:

* any chronic cardiovascular condition or metabolic condition
* kidney disease
* gastro-intestinal disease
* milk or dairy protein allergies
* lactose intolerance
* chronic lung conditions
* any condition that could potentially prevent participant from performing exercise
* allergy to local anaesthetics
* cumulative x-ray exposure and cumulative muscle biopsies

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Body composition | 12 weeks
Bone mineral density | 12 weeks
VO2 peak | 12 weeks

SECONDARY OUTCOMES:
mitochondrial enzyme activity | 12 weeks
muscle oxidative stress | 12 weeks
muscle capillary density | 12 weeks
blood lipids | 12 weeks
blood inflammatory markers | 12 weeks
blood markers of bone turnover | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Roy, PhD, Principal Investigator — Brock University
Locations (1):
- Brock University, St. Catharines, Ontario, Canada

REFERENCES:
- See also: University website — http://www.brocku.ca
- See also: Sponsor of the trial — http://www.dairyfarmers.ca/